CLINICAL TRIAL: NCT04331067
Title: Phase Ib/II Study to Evaluate Safety and Tolerability of Neoadjuvant Nivolumab and Chemotherapy in Patients With Localized Triple-negative Breast Cancer
Brief Title: Neoadjuvant Nivolumab and Chemotherapy in Patients With Localized Triple-negative Breast Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202007016
Record Dates: First submitted 2020-03-30; First posted 2020-04-02 (Actual); Results first posted 2024-05-16 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Paclitaxel; Carboplatin; Nivolumab; cabiralizumab; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm A: Neoadjuvant chemo + nivolumab (Active Comparator): -Neoadjuvant chemotherapy consists of paclitaxel and carboplatin. Paclitaxel will be given intravenously (IV) at a dose of 80 mg/m^2 on a weekly basis for 12 weeks. Carboplatin will be given IV at a dose of AUC 5 every 3 weeks for 12 weeks. Nivolumab will be given IV at a dose of 240 mg every 2 weeks for 12 weeks. Nivolumab will be administered first, followed by carboplatin, followed by paclitaxel.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Biological: Nivolumab; Procedure: Tumor biopsy; Procedure: Bone marrow; Procedure: Blood draw
- Arm B: Neoadjuvant chemo + nivolumab + cabiralizumab (Experimental): As of Amendment #7 IRB approved 10/13/2022: The study will no longer enroll to Arm B. Cabiralizumab will no longer be given.
  * Neoadjuvant chemotherapy consists of paclitaxel and carboplatin. Paclitaxel will be given intravenously (IV) at a dose of 80 mg/m^2 on a weekly basis for 12 weeks. Carboplatin will be given IV at a dose of AUC 5 every 3 weeks for 12 weeks. Nivolumab will be given IV at a dose of 240 mg every 2 weeks for 12 weeks. Nivolumab will be administered first, followed by carboplatin, followed by paclitaxel.
  * Cabiralizumab will be given IV at a dose of 4 mg/kg every 2 weeks for 12 weeks.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Biological: Nivolumab; Biological: Cabiralizumab; Procedure: Tumor biopsy; Procedure: Bone marrow; Procedure: Blood draw
- Unrandomized Arm: Neoadjuvant Chemo + Nivolumab (Experimental): * As of Amendment #7 IRB approved 10/13/2022: The study will no longer enroll to Arm B. Cabiralizumab will no longer be given. Remaining patients will be enrolled in single arm study.
  * Neoadjuvant chemotherapy consists of paclitaxel and carboplatin. Paclitaxel will be given intravenously (IV) at a dose of 80 mg/m^2 on a weekly basis for 12 weeks. Carboplatin will be given IV at a dose of AUC 5 every 3 weeks for 12 weeks. Nivolumab will be given IV at a dose of 240 mg every 2 weeks for 12 weeks. Nivolumab will be administered first, followed by carboplatin, followed by paclitaxel.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Biological: Nivolumab; Procedure: Tumor biopsy; Procedure: Bone marrow; Procedure: Blood draw

INTERVENTIONS:
Drug: Paclitaxel — -Given standard of care
  Other Names: Taxol
Drug: Carboplatin — -Given standard of care
  Other Names: Paraplatin
Biological: Nivolumab — -Given standard of care
  Other Names: Opdivo; BMS-936558
Biological: Cabiralizumab — -Will be provided by Bristol Myers Squibb
  Other Names: BMS-986227
  Arms: Arm B: Neoadjuvant chemo + nivolumab + cabiralizumab
Procedure: Tumor biopsy — -Baseline, week 5, surgery, and at time of relapse (optional)
Procedure: Bone marrow — -Time of port placement (baseline), time of surgery, and time of recurrence (optional)
Procedure: Blood draw — -Baseline, week 5, prior to surgery , post-surgery follow-up (typically 3-4 weeks post-surgery), and disease progression (optional)

SUMMARY:
Prior to Amendment #7: The hypothesis of this study is that the combination of cabiralizumab and nivolumab with neoadjuvant chemotherapy will decrease tumor associated macrophages (TAMs) and increase tumor infiltrating lymphocytes (TIL) compared to neoadjuvant chemotherapy plus nivolumab in patients with early stage triple-negative breast cancer (TNBC) and improve clinical outcomes.

As of Amendment #7 IRB approved 10/13/2022: The study will no longer enroll to Arm B. Cabiralizumab will no longer be given. The hypothesis of this study is that on-treatment tumor associated macrophages (TAMs) and tumor infiltrating lymphocytes (TILs) will improve (reduced TAMs, increased TILs) following neoadjuvant nivolumab with chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed newly diagnosed ER-/HER2- breast cancer. ER and PR < Allred score of 3 or < 1% positive staining cells in the invasive component of the tumor. HER2 negative by FISH or IHC staining 0 or 1+ according to NCCN guidelines.
* Clinical stage II or III (by AJCC 8th edition at least T2, any N, M0 or if N+ then any T) breast cancer eligible for neoadjuvant chemotherapy with complete surgical excision of the breast cancer after neoadjuvant therapy as the treatment goal.
* Tumor size at least 2 cm in one dimension by clinical or radiographic exam (WHO criteria). Patients with histologically confirmed or clinically palpable lymph nodes may be enrolled regardless of tumor size. A palpable mass is not required as long as the mass is at least 2 cm in one dimension by radiographic exam. 2D measurements should be completed during screening if available.
* No prior therapy for this disease
* At least 18 years of age.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
* Normal bone marrow and organ function as defined below:

  * Leukocytes ≥ 2,000/mcL (stable off any growth factor within 4 weeks of first study treatment administration)
  * Absolute neutrophil count ≥ 1,500/mcL (stable off any growth factor within 4 weeks of first study treatment administration)
  * Platelets ≥ 100,000/mcL (stable off any growth factor within 4 weeks of first study treatment administration)
  * Hemoglobin ≥8.5 g/dl (transfusion to achieve this level is not permitted within 2 weeks of first study treatment administration)
  * Total bilirubin ≤ 1.5 x institutional upper limit of normal (IULN) (except participants with Gilbert's Syndrome who must have normal direct bilirubin)
  * AST(SGOT)/ALT(SGPT) ≤ 2.0 x IULN
  * Alkaline phosphatase <2.5 x ULN
  * Serum creatinine < 1.5 x ULN or creatinine clearance > 40 mL/min by Cockcroft-Gault
  * Albumin ≥ 3 g/dL
  * INR and aPTT <1.5 x IULN (This applies only to patients who do not receive therapeutic anticoagulation; patients receiving therapeutic anticoagulation, such as low-molecular-weight heparin or warfarin, should be on a stable dose).
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of study treatment.
* Women must not be breastfeeding.
* WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study treatment(s) and for a total of 5 months post-treatment completion.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).
* Consent for fresh pre-treatment, on-treatment, biopsy samples at acceptable clinical risk, as judged by the investigator.
* Participants must be willing and able to comply with scheduled visits, treatment schedule, and laboratory testing

Exclusion Criteria:

* Prior treatment with immunotherapy for cancer
* Known metastatic disease
* Known invasive cancer in contralateral breast
* Patients with a previous history of non-breast malignancy are eligible only if they meet the following criteria for a cancer survivor:

  * Has undergone potentially curative therapy for all prior malignancies AND
  * Has been considered disease-free for at least 1 year (with the exception of basal cell or squamous cell carcinoma of the skin or carcinoma-in-situ of the cervix.
* Currently receiving any other investigational agents.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to paclitaxel, carboplatin, nivolumab, or other agents used in the study. Patients who have received multiple blood transfusions.
* Evidence of uncontrolled ongoing or active infection, requiring parenteral anti-bacterial, anti-viral, or anti-fungal therapy ≤ 7 days prior to administration of study treatment. Patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or chronic obstructive pulmonary disease) are eligible.
* Patients with prior allogeneic bone marrow transplantation or prior solid organ transplantation.
* History or risk of autoimmune disease, including, but not limited to, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease (Crohn's disease and ulcerative colitis), vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Bell's palsy, Guillain-Barré syndrome, multiple sclerosis, autoimmune thyroid disease, vasculitis, or glomerulonephritis.

  * Patients with a history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone may be eligible.
  * Patients with controlled Type 1 diabetes mellitus on a stable insulin regimen may be eligible.
  * Patients with eczema, psoriasis, lichen simplex chronicus of vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are permitted provided that they meet the following conditions:

    * Patients with psoriasis must have a baseline ophthalmologic exam to rule out ocular manifestations
    * Rash must cover less than 10% of body surface area (BSA)
    * Disease is well controlled at baseline and only requiring low potency topical steroids (e.g., hydrocortisone 2.5%, hydrocortisone butyrate 0.1%, flucinolone 0.01%, desonide 0.05%, aclometasone dipropionate 0.05%)
    * No acute exacerbations of underlying condition within the last 12 months (not requiring psoralen plus ultraviolet A radiation [PUVA], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors; high potency or oral steroids)
* History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest computed tomography (CT) scan.
* Uncontrolled or significant cardiovascular disease
* History of any chronic hepatitis as evidenced by the following:

  * Positive test for hepatitis B surface antigen
  * Positive test for qualitative hepatitis C viral load (by polymerase chain reaction [PCR]).
* Positive test for latent tuberculosis (TB) at screening (e.g. T-SPOT or Quantiferon test) or evidence of active TB.
* Major surgical procedure within 28 days prior to Cycle 1, Day 1 or anticipation of need for a major surgical procedure during the course of the study with the exception of the planned breast cancer surgery that is part of the trial design. Participants must have recovered from the effects of major surgery or significant traumatic injury at least 14 days before the first dose of study treatment.
* Any uncontrolled medical condition which, in the opinion of the Investigator, would pose a risk to participant safety or interfere with study participation or interpretation of individual participant results.
* Treatment with systemic immunosuppressive medications (including, but not limited to, prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 2 weeks prior to Cycle 1, Day 1.

  * Patients who have received acute, low dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled.
  * The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension or adrenocortical insufficiency is allowed. The use of replacement doses of prednisone or other corticosteroid for adrenocortical insufficiency is allowed
  * Participants with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of start of study treatment. Inhaled or topical steroids and adrenal replacement steroid doses > 10 mg daily prednisone equivalent are permitted in the absence of active autoimmune disease.
* Evidence of coagulopathy or bleeding diathesis.
* Ascites needing paracentesis or medical management.
* Patients positive for human immunodeficiency virus (HIV) are NOT excluded from this study, but HIV-positive patients must have:

  * A stable regimen of highly active anti-retroviral therapy (HAART)
  * No requirement for concurrent antibiotics or antifungal agents for the prevention of opportunistic infections
  * A CD4 count above 250 cells/mcL and an undetectable HIV viral load on standard PCR-based tests

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2026-05-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Davis, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A: Neoadjuvant Chemo + Nivolumab | Arm B: Neoadjuvant Chemo + Nivolumab + Cabiralizumab | Unrandomized Arm: Neoadjuvant Chemo + Nivolumab
Started | 6 | 6 | 3
Completed | 4 | 3 | 2
Not Completed | 2 | 3 | 1
Not completed — Adverse Event | 1 | 3 | 1
Not completed — Physician decision - patient not compliant with visits | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Neoadjuvant Chemo + Nivolumab | Arm B: Neoadjuvant Chemo + Nivolumab + Cabiralizumab | Unrandomized Arm: Neoadjuvant Chemo + Nivolumab | Total
Number analyzed (Participants) | 6 | 6 | 3 | 15
Age, Continuous [Median (Full Range); unit: years] | 55 [46 to 63] | 55.5 [38 to 68] | 62 [53 to 63] | 57 [38 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 3 | 15
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 6 | 5 | 3 | 14
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 2 | 6
  White | 4 | 4 | 1 | 9
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 3 | 15

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Tumor Infiltrating Lymphocytes (TILs)
Description: -Stromal TIL score is defined as the percentage of tumor stroma area that was occupied by mononuclear inflammatory cells.
Time Frame: Baseline and week 5
Population: Arm A and Unrandomized Arm were analyzed together as the treatment received was the same. There were 2 participants with missing data in Arm A/Unrandomized Arm and 2 participants with missing data in Arm B and these participants were not included in the analysis.
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Arm A and Unrandomized Arm: Neoadjuvant Chemo + Nivolumab: -Neoadjuvant chemotherapy consists of paclitaxel and carboplatin. Paclitaxel will be given intravenously (IV) at a dose of 80 mg/m^2 on a weekly basis for 12 weeks. Carboplatin will be given IV at a dose of AUC 5 every 3 weeks for 12 weeks. Nivolumab will be given IV at a dose of 240 mg every 2 weeks for 12 weeks. Nivolumab will be administered first, followed by carboplatin, followed by paclitaxel.
Arm/Group | Arm A and Unrandomized Arm: Neoadjuvant Chemo + Nivolumab | Arm B: Neoadjuvant Chemo + Nivolumab + Cabiralizumab
Number analyzed (Participants) | 7 | 4
percent change | 95.2 (121) | 1.63 (82.5)

2. Primary Outcome: Percent Change in Tumor Associated Macrophages (TAMs)
Time Frame: Baseline and week 5
Population: Arm A and Unrandomized Arm were analyzed together as the treatment received was the same. There were 3 participants with missing data in Arm A/Unrandomized Arm and 3 participants with missing data in Arm B and these participants were not included in the analysis.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Arm A and Unrandomized Arm: Neoadjuvant Chemo + Nivolumab | Arm B: Neoadjuvant Chemo + Nivolumab + Cabiralizumab
Number analyzed (Participants) | 6 | 3
percent change | 31.8 (32.1) | -38.7 (63.6)

3. Primary Outcome: Safety of the Regimen as Measured by Incidence of Adverse Events (Safety lead-in Only)
Description: Safety lead-in consists of the first 12 patients treated on the study (Arm A and Arm B).
Time Frame: From start of treatment through 100 days after last day of study treatment or surgery whichever occurs first (approximately 16 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Neoadjuvant Chemo + Nivolumab | Arm B: Neoadjuvant Chemo + Nivolumab + Cabiralizumab
Number analyzed (Participants) | 6 | 6
Participants
  Grade 1-2 anemia | 4 | 2
  Grade 3-4 anemia | 2 | 4
  Grade 1-2 lymph node pain | 1 | 0
  Grade 1-2 supraventricular tachycardia | 0 | 1
  Grade 1-2 adrenal insufficiency | 1 | 0
  Grade 1-2 diabetes | 1 | 0
  Grade 1-2 hypoparathyroidism | 0 | 1
  Grade 1-2 hypothyroidism | 1 | 0
  Grade 1-2 blurred vision | 1 | 1
  Grade 1-2 eye pain | 0 | 1
  Grade 1-2 periorbital edema | 0 | 3
  Grade 3-4 periorbital edema | 0 | 1
  Grade 1-2 photophobia | 0 | 1
  Grade 3-4 uveitis | 0 | 1
  Grade 1-2 watering eyes | 0 | 3
  Grade 1-2 abdominal pain | 2 | 0
  Grade 1-2 constipation | 2 | 1
  Grade 1-2 diarrhea | 2 | 3
  Grade 1-2 dry mouth | 0 | 2
  Grade 1-2 dyspepsia | 2 | 1
  Grade 1-2 dysphagia | 0 | 1
  Grade 1-2 gastroesophageal reflux disease | 1 | 0
  Grade 1-2 gas pain | 0 | 1
  Grade 1-2 gastrointestinal pain | 1 | 0
  Grade 1-2 mucositis oral | 0 | 5
  Grade 1-2 nausea | 5 | 5
  Grade 1-2 vomiting | 2 | 1
  Grade 3-4 vomiting | 0 | 1
  Grade 1-2 chills | 2 | 0
  Grade 1-2 edema limbs | 1 | 3
  Grade 1-2 edema trunk | 1 | 0
  Grade 1-2 fatigue | 6 | 4
  Grade 1-2 fever | 1 | 3
  Grade 1-2 flu like symptoms | 0 | 1
  Grade 1-2 generalized body aches | 1 | 0
  Grade 1-2 localized edema | 0 | 1
  Grade 1-2 neck edema | 0 | 1
  Grade 1-2 non-cardiac chest pain | 3 | 0
  Grade 1-2 allergic reaction | 0 | 1
  Grade 1-2 bronchitis | 0 | 1
  Grade 1-2 cold symptoms | 0 | 1
  Grade 1-2 conjunctivitis | 0 | 1
  Grade 1-2 eye infection | 0 | 1
  Grade 1-2 folliculitis | 1 | 0
  Grade 3-4 sepsis | 1 | 0
  Grade 1-2 thrush | 1 | 1
  Grade 3-4 thrush | 0 | 1
  Grade 1-2 urinary tract infection | 0 | 1
  Grade 1-2 fall | 1 | 0
  Grade 1-2 infusion related reaction | 1 | 2
  Grade 1-2 seroma | 1 | 0
  Grade 1-2 alanine aminotransferase increased | 4 | 6
  Grade 1-2 alkaline phosphtase increased | 3 | 5
  Grade 1-2 aspartate aminotransferase increased | 1 | 4
  Grade 3-4 aspartate aminotransferase increased | 0 | 2
  Grade 1-2 blood lactate dehydrogenase increased | 4 | 6
  Grade 1-2 cardiac troponin I increased | 0 | 2
  Grade 1-2 cardiac troponin T increased | 0 | 1
  Grade 1-2 cholesterol high | 1 | 0
  Grade 1-2 CPK increased | 0 | 2
  Grade 3-4 CPK increased | 0 | 4
  Grade 1-2 creatinine increased | 1 | 1
  Grade 3-4 creatinine increased | 0 | 1
  Grade 1-2 fibrinogen decreased | 0 | 1
  Grade 1-2 haptoglobin decreased | 0 | 1
  Grade 1-2 INR increased | 0 | 2
  Grade 1-2 lipase increased | 1 | 5
  Grade 1-2 lymphocyte count decreased | 2 | 1
  Grade 3-4 lymphocyte count decreased | 1 | 4
  Grade 1-2 neutrophil count decreased | 2 | 3
  Grade 3-4 neutrophil count decreased | 2 | 3
  Grade 1-2 platelet count decreased | 3 | 4
  Grade 3-4 platelet count decreased | 1 | 2
  Grade 1-2 thyroid stimulating hormone increased | 1 | 2
  Grade 3-4 weight gain | 0 | 1
  Grade 1-2 weight loss | 0 | 1
  Grade 3-4 weight loss | 0 | 1
  Grade 1-2 white blood cell decreased | 3 | 3
  Grade 3-4 white blood cell decreased | 2 | 3
  Grade 1-2 anorexia | 1 | 3
  Grade 1-2 dehydration | 1 | 1
  Grade 3-4 dehydration | 0 | 1
  Grade 1-2 hypercalcemia | 1 | 1
  Grade 1-2 hyperglycemia | 2 | 3
  Grade 1-2 hyperkalemia | 1 | 0
  Grade 1-2 hypernatremia | 0 | 1
  Grade 3-4 hypernatremia | 0 | 1
  Grade 1-2 hypertriglyceridemia | 1 | 2
  Grade 1-2 hyperuricemia | 0 | 2
  Grade 1-2 hypoalbuminemia | 1 | 2
  Grade 1-2 hypocalcemia | 1 | 1
  Grade 3-4 hypocalcemia | 0 | 2
  Grade 1-2 hypoglycemia | 0 | 2
  Grade 1-2 hypokalemia | 1 | 1
  Grade 3-4 hypokalemia | 0 | 2
  Grade 1-2 hypomagnesemia | 0 | 1
  Grade 3-4 hypomagnesemia | 0 | 1
  Grade 1-2 hyponatremia | 2 | 2
  Grade 1-2 hypophosphatemia | 0 | 3
  Grade 1-2 arthralgia | 0 | 1
  Grade 1-2 arthritis | 1 | 0
  Grade 1-2 back aches | 1 | 0
  Grade 1-2 back pain | 0 | 1
  Grade 1-2 back spasms | 1 | 0
  Grade 1-2 bilateral rib pain | 1 | 0
  Grade 1-2 bone pain | 2 | 2
  Grade 3-4 bone pain | 0 | 1
  Grade 1-2 generalized muscle weakness | 2 | 1
  Grade 3-4 generalized muscle weakness | 0 | 1
  Grade 1-2 muscle cramp | 0 | 1
  Grade 1-2 muscle soreness | 1 | 0
  Grade 1-2 myalgia | 1 | 2
  Grade 3-4 myositis | 0 | 2
  Grade 1-2 rhabdomyolysis | 0 | 1
  Grade 1-2 shoulder pain | 1 | 0
  Grade 1-2 dizziness | 4 | 4
  Grade 1-2 dysgeusia | 2 | 3
  Grade 1-2 encephalopathy | 0 | 1
  Grade 1-2 headache | 4 | 2
  Grade 1-2 jitters | 1 | 0
  Grade 1-2 memory impairment | 1 | 0
  Grade 1-2 peripheral motor neuropathy | 1 | 1
  Grade 1-2 peripheral sensory neuropathy | 2 | 5
  Grade 3-4 peripheral sensory neuropathy | 1 | 0
  Grade 3-4 syncope | 1 | 0
  Grade 1-2 tremors | 0 | 1
  Grade 1-2 agitation | 2 | 0
  Grade 1-2 altered mental state | 0 | 1
  Grade 1-2 depression | 2 | 0
  Grade 1-2 insomnia | 2 | 3
  Grade 1-2 mania | 1 | 0
  Grade 3-4 acute kidney injury | 0 | 1
  Grade 1-2 glucosuria | 3 | 3
  Grade 1-2 hematuria | 1 | 3
  Grade 1-2 proteinuria | 1 | 3
  Grade 1-2 urinary urgency | 1 | 0
  Grade 1-2 areola pain | 0 | 1
  Grade 1-2 breast edema | 0 | 1
  Grade 1-2 breast pain | 1 | 1
  grade 1-2 irregular menstruation | 0 | 1
  Grade 1-2 allergic rhinitis | 1 | 0
  Grade 1-2 cough | 2 | 2
  Grade 1-2 dyspnea | 4 | 1
  Grade 1-2 epistaxis | 3 | 3
  Grade 1-2 productive cough | 1 | 0
  Grade 1-2 sore throat | 0 | 1
  Grade 1-2 alopecia | 4 | 4
  Grade 1-2 dermatitis radiation | 1 | 0
  Grade 1-2 dry skin | 0 | 1
  Grade 1-2 flat, lacy rash | 0 | 1
  Grade 1-2 hyperhidrosis | 1 | 0
  Grade 1-2 macular rash | 1 | 0
  Grade 1-2 palmar-plantar erythrodysesthesia syndrome | 1 | 0
  Grade 1-2 photosensitivity | 0 | 1
  Grade 1-2 pruritus | 1 | 2
  Grade 1-2 rash acneiform | 0 | 1
  Grade 1-2 rash maculo-papular | 3 | 4
  Grade 1-2 skin pain on chest and arms | 0 | 1
  Grade 3-4 skin ulceration | 0 | 2
  Grade 1-2 hot flashes | 2 | 0
  Grade 1-2 hypertension | 1 | 1
  Grade 3-4 hypertension | 2 | 3
  Grade 1-2 hypotension | 1 | 1
  Grade 3-4 hypotension | 1 | 0
  Grade 1-2 thromboembolic event | 2 | 1
  Grade 3-4 thromboembolic event | 1 | 0

4. Secondary Outcome: Pathological Complete Response (pCR)
Description: -A pathologic complete response (pCR) is defined as no histology evidence of invasive tumor cells in the surgical breast specimen and sentinel or axillary lymph nodes.
Time Frame: At time of surgery (average of 12 weeks)
Population: 1 participant in Arm A and 1 participant in Arm B did not have surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Neoadjuvant Chemo + Nivolumab | Arm B: Neoadjuvant Chemo + Nivolumab + Cabiralizumab | Unrandomized Arm: Neoadjuvant Chemo + Nivolumab
Number analyzed (Participants) | 5 | 5 | 3
Participants | 3 | 2 | 2

5. Secondary Outcome: Recurrence-free Survival (RFS)
Description: -RFS is defined from time of surgery to the earliest time of recurrence, time to development of a second cancer, or time to death from any cause.
Time Frame: Through completion of follow-up (estimated to be 3 years and 12 weeks)
Reporting Status: Not Posted

6. Secondary Outcome: Adverse Events Measured by Number of Participants With Nivolumab Related Grade 3 or Higher Adverse Events
Description: Treatment related means either possibly, probably, or definitely related to nivolumab
Time Frame: From start of treatment through 100 days after last infusion of study treatment or surgery whichever occurs first (approximately 16 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Neoadjuvant Chemo + Nivolumab | Arm B: Neoadjuvant Chemo + Nivolumab + Cabiralizumab | Unrandomized Arm: Neoadjuvant Chemo + Nivolumab
Number analyzed (Participants) | 6 | 6 | 3
Participants
  Anemia | 1 | 1 | 1
  Thrush | 0 | 1 | 0
  Aspartate aminotransferase increased | 0 | 2 | 0
  CPK increased | 0 | 3 | 0
  Creatinine increased | 0 | 1 | 0
  Lymphocyte count decreased | 0 | 1 | 0
  Neutrophil count decreased | 0 | 1 | 0
  Platelet count decreased | 0 | 2 | 0
  Weight gain | 0 | 1 | 0
  Dehydration | 0 | 1 | 0
  Hypocalcemia | 0 | 1 | 0
  Hypokalemia | 0 | 1 | 1
  Generalized muscle weakness | 0 | 1 | 0
  Myositis | 0 | 2 | 0
  Acute kidney injury | 0 | 1 | 0

7. Secondary Outcome: Adverse Events Measured by Number of Participants With Carboplain Related Grade 3 or Higher Adverse Events
Description: Treatment related means either possibly, probably, or definitely related to carboplatin
Time Frame: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Neoadjuvant Chemo + Nivolumab | Arm B: Neoadjuvant Chemo + Nivolumab + Cabiralizumab | Unrandomized Arm: Neoadjuvant Chemo + Nivolumab
Number analyzed (Participants) | 6 | 6 | 3
Participants
  Anemia | 2 | 2 | 1
  Sepsis | 1 | 0 | 0
  Thrush | 0 | 1 | 0
  Aspartate aminotransferase increased | 0 | 1 | 0
  Lymphocyte count decreased | 0 | 2 | 0
  Neutrophil count decreased | 1 | 1 | 0
  Platelet count decreased | 1 | 1 | 0
  White blood cell decreased | 1 | 1 | 0
  Dehydration | 0 | 1 | 0
  Hypernatremia | 0 | 1 | 0
  Hypocalcemia | 0 | 1 | 0
  Hypokalemia | 0 | 1 | 1
  Hypomagnesemia | 0 | 1 | 0
  Peripheral sensory neuropathy | 1 | 0 | 0
  Acute kidney injury | 0 | 1 | 0
  Hypotension | 1 | 0 | 0

8. Secondary Outcome: Adverse Events Measured by Number of Participants With Paclitaxel Related Grade 3 or Higher Adverse Events
Description: Treatment related means either possibly, probably, or definitely related to paclitaxel
Time Frame: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Neoadjuvant Chemo + Nivolumab | Arm B: Neoadjuvant Chemo + Nivolumab + Cabiralizumab | Unrandomized Arm: Neoadjuvant Chemo + Nivolumab
Number analyzed (Participants) | 6 | 6 | 3
Participants
  Anemia | 2 | 2 | 1
  Sepsis | 1 | 0 | 0
  Thrush | 0 | 1 | 0
  Aspartate aminotransferase increased | 0 | 1 | 0
  Lymphocyte count decreased | 0 | 2 | 0
  Neutrophil count decreased | 1 | 2 | 0
  Platelet count decreased | 1 | 1 | 0
  Weight gain | 0 | 1 | 0
  White blood cell decreased | 1 | 2 | 0
  Dehydration | 0 | 1 | 0
  Hypernatremia | 0 | 1 | 0
  Hypocalcemia | 0 | 1 | 0
  Hypokalemia | 0 | 1 | 1
  Hypomagnesemia | 0 | 1 | 0
  Peripheral sensory neuropathy | 1 | 0 | 0
  Acute kidney injury | 0 | 1 | 0
  Hypotension | 1 | 0 | 0

9. Secondary Outcome: Adverse Events Measured by Number of Participants With Cabiralizumab Related Grade 3 or Higher Adverse Events
Description: Treatment related means either possibly, probably, or definitely related to cabiralizumab
Time Frame: as for outcome 6
Population: This outcome measure is only for Arm B as that arm is the only arm that received cabiralizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Neoadjuvant Chemo + Nivolumab | Arm B: Neoadjuvant Chemo + Nivolumab + Cabiralizumab | Unrandomized Arm: Neoadjuvant Chemo + Nivolumab
Number analyzed (Participants) | 0 | 6 | 0
Participants
  Anemia |  | 1 |
  Periorbital edema |  | 1 |
  Uveitis |  | 1 |
  Thrush |  | 1 |
  Aspartate aminotransferase increased |  | 2 |
  CPK increased |  | 4 |
  Lymphocyte count decreased |  | 1 |
  Neutrophil count decreased |  | 1 |
  Platelet count decreased |  | 2 |
  Weight gain |  | 1 |
  Dehydration |  | 1 |
  Hypocalcemia |  | 1 |
  Hypokalemia |  | 1 |
  Generalized muscle weakness |  | 1 |
  Myositis |  | 2 |
  Acute kidney injury |  | 1 |

10. Secondary Outcome: Compare the Percent Change of Tumor Associated Macrophages (TAMs) Between Participants Who Achieve pCR Versus Those Who do Not
Description: as for outcome 4
Time Frame: At time of surgery (average of 12 weeks)
Population: Arm A and Unrandomized Arm were analyzed together as the treatment received was the same. There were 2 participants with missing data in Arm A/Unrandomized Arm and 3 participants with missing data in Arm B and these participants were not included in the analysis.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Arm A and Unrandomized Arm: Neoadjuvant Chemo + Nivolumab | Arm B: Neoadjuvant Chemo + Nivolumab + Cabiralizumab
Number analyzed (Participants) | 7 | 3
percent change
  non-pCR: number analyzed (Participants) | 4 | 1
  non-pCR | 41.9 (92.1) | 82.8 (NA) — There is no standard deviation as there is only data for one participant.
  pCR: number analyzed (Participants) | 3 | 2
  pCR | 166 (134) | -19.9 (107)

11. Secondary Outcome: Compare the Percent Change of Tumor Infiltrating Lymphocytes (TILs) Between Participants Who Achieve pCR Versus Those Who do Not
Description: * Stromal TIL score is defined as the percentage of tumor stroma area that was occupied by mononuclear inflammatory cells.
  * A pathologic complete response (pCR) is defined as no histology evidence of invasive tumor cells in the surgical breast specimen and sentinel or axillary lymph nodes.
Time Frame: At time of surgery (average of 12 weeks)
Population: Arm A and Unrandomized Arm were analyzed together as the treatment received was the same. There were 3 participants with missing data in Arm A/Unrandomized Arm and 4 participants with missing data in Arm B and these participants were not included in the analysis.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Arm A and Unrandomized Arm: Neoadjuvant Chemo + Nivolumab | Arm B: Neoadjuvant Chemo + Nivolumab + Cabiralizumab
Number analyzed (Participants) | 6 | 2
percent change
  non-pCR: number analyzed (Participants) | 3 | 1
  non-pCR | 11.1 (19.9) | 32.2 (NA) — There is no standard deviation as there is only data for one participant.
  pCR: number analyzed (Participants) | 3 | 1
  pCR | 52.5 (29.9) | -90.6 (NA) — There is no standard deviation as there is only data for one participant.

ADVERSE EVENTS:
Time Frame: Adverse events were collected from start of treatment through 100 days after last treatment or day of surgery, whichever was first. All-cause mortality was collected from start of treatment through completion of follow-up (up to 36 months).
Arm/Group | Arm A: Neoadjuvant Chemo + Nivolumab | Arm B: Neoadjuvant Chemo + Nivolumab + Cabiralizumab | Unrandomized Arm: Neoadjuvant Chemo + Nivolumab
All-Cause Mortality (participants affected / at risk) | 1/6 | 1/6 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/6 | 3/6 | 0/3
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Neoadjuvant Chemo + Nivolumab (N=6) | Arm B: Neoadjuvant Chemo + Nivolumab + Cabiralizumab (N=6) | Unrandomized Arm: Neoadjuvant Chemo + Nivolumab (N=3)
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Thromboembolic event (Vascular disorders) | 1 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Neoadjuvant Chemo + Nivolumab (N=6) | Arm B: Neoadjuvant Chemo + Nivolumab + Cabiralizumab (N=6) | Unrandomized Arm: Neoadjuvant Chemo + Nivolumab (N=3)
Anemia (Blood and lymphatic system disorders) | 6 | 5 | 3
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 1
Diabetes (Endocrine disorders) | 1 | 0 | 0
Hypoparathyroidism (Endocrine disorders) | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0
Blurred vision (Eye disorders) | 1 | 1 | 0
Eye pain (Eye disorders) | 0 | 1 | 0
Periorbital edema (Eye disorders) | 0 | 4 | 0
Photophobia (Eye disorders) | 0 | 1 | 0
Uveitis (Eye disorders) | 0 | 1 | 0
Watering eyes (Eye disorders) | 0 | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 1 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 3 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0
Gas pain (Gastrointestinal disorders) | 0 | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 5 | 1
Nausea (Gastrointestinal disorders) | 5 | 5 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1 | 0
Chills (General disorders) | 2 | 0 | 0
Edema limbs (General disorders) | 1 | 3 | 0
Edema trunk (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 6 | 4 | 3
Fever (General disorders) | 1 | 3 | 0
Flu like symptoms (General disorders) | 0 | 1 | 0
Generalized body aches (General disorders) | 1 | 0 | 0
Localized edema (General disorders) | 0 | 1 | 0
Neck edema (General disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 3 | 0 | 0
Pain (General disorders) | 0 | 0 | 2
Allergic reaction (Immune system disorders) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
Cold symptoms (Infections and infestations) | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 0
Eye infection (Infections and infestations) | 0 | 1 | 1
Folliculitis (Infections and infestations) | 1 | 0 | 1
Paronychia (Infections and infestations) | 0 | 0 | 1
Thrush (Infections and infestations) | 1 | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 2 | 0
Seroma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 4 | 6 | 1
Alkaline phosphatase increased (Investigations) | 3 | 5 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 6 | 1
Blood lactate dehydrogenase increased (Investigations) | 4 | 6 | 0
CPK increased (Investigations) | 0 | 6 | 0
Cardiac troponin I increased (Investigations) | 0 | 2 | 0
Cardiac troponin T increased (Investigations) | 0 | 1 | 0
Cholesterol high (Investigations) | 1 | 0 | 0
Creatinine increased (Investigations) | 1 | 2 | 0
Fibrinogen decreased (Investigations) | 0 | 1 | 0
Haptoglobin decreased (Investigations) | 0 | 1 | 0
INR increased (Investigations) | 0 | 2 | 0
Lipase increased (Investigations) | 1 | 5 | 0
Lymphocyte count decreased (Investigations) | 3 | 5 | 2
Lymphocyte count increased (Investigations) | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 3 | 6 | 3
Platelet count decreased (Investigations) | 4 | 5 | 1
Thyroid stimulating hormone increased (Investigations) | 1 | 2 | 0
Weight gain (Investigations) | 0 | 1 | 0
Weight loss (Investigations) | 0 | 2 | 1
White blood cell count decreased (Investigations) | 5 | 6 | 3
Anorexia (Metabolism and nutrition disorders) | 1 | 3 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 3 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypernatremia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 2 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 2 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 3 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 3 | 1
Hypomagenesemia (Metabolism and nutrition disorders) | 0 | 2 | 1
Hyponatremia (Metabolism and nutrition disorders) | 2 | 2 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back aches (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bilateral rib pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle soreness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 4 | 4 | 1
Dysgeusia (Nervous system disorders) | 2 | 3 | 2
Encephalopathy (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 4 | 2 | 2
Jitters (Nervous system disorders) | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 1 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 5 | 3
Syncope (Nervous system disorders) | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0
Agitation (Psychiatric disorders) | 2 | 0 | 0
Altered mental state (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 2 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 3 | 1
Mania (Psychiatric disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0
Glucosuria (Renal and urinary disorders) | 3 | 3 | 0
Hematuria (Renal and urinary disorders) | 1 | 3 | 0
Proteinuria (Renal and urinary disorders) | 1 | 3 | 1
Urinary urgency (Renal and urinary disorders) | 1 | 0 | 0
Areola pain (Reproductive system and breast disorders) | 0 | 1 | 0
Breast edema (Reproductive system and breast disorders) | 0 | 1 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 1 | 0
Irregular menstruation (Reproductive system and breast disorders) | 0 | 1 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 4 | 2
Dermatitis radiation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Flat, lacy rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hyperhydrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Macular rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 3 | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin pain on chest and arms (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Hot flashes (Vascular disorders) | 2 | 0 | 1
Hypertension (Vascular disorders) | 3 | 4 | 0
Hypotension (Vascular disorders) | 2 | 1 | 0
Thromboembolic event (Vascular disorders) | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-27): https://cdn.clinicaltrials.gov/large-docs/67/NCT04331067/Prot_SAP_000.pdf